CLINICAL TRIAL: NCT04172818
Title: Feasibility Study of a Diary for Allogenic Hematopoietic Stem Cell Transplantation Patients and Families
Acronym: JACintHE
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Centre Hospitalier Universitaire, Amiens (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: PI2019_843_0005
Record Dates: First submitted 2019-11-14; First posted 2019-11-21 (Actual); Last update posted 2023-03-22 (Actual); Status verified 2023-03

CONDITIONS: Hematopoietic/Lymphoid Cancer; Psychological Disorder
Keywords: allogenic hematopoietic stem cell transplantation; diary; psychological disorders
MeSH Terms: conditions — Hematologic Neoplasms; Mental Disorders

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Patients with diary (Experimental): Evaluation the psychological impact of a diary on the patients hospitalized for allogenic hematopoetic stem cell transplantation and on their relatives.
  Interventions: Behavioral: quality of life questionnaire

INTERVENTIONS:
Behavioral: quality of life questionnaire — Since 10 years ago, diaries are used in intensive care unit to limit these symptoms after a coma.In analogy, the diary for patients with allogenic hematopoietic stem cell transplantation could be a mean to reduce the psychological adverse impact and long term consequences. The psychological impact of a diary on patients hospitalized for allogenic hematopoetic stem cell transplantation and on their relatives will be evaluated.

SUMMARY:
Allogenic hematopoietic stem cell transplantation is a specific time during hematological disease management for the patients, theirs relatives and the healthcare team. This heavy treatment is most of the time the last possible curative therapy and could cause many side effects such as infectious diseases and graft versus host reaction. The protective isolation is also a source of physical and psychological isolation. Published studies reported depressive syndrome, anxiety symptoms and post-traumatic stress disorders for patients and their families. Since 10 years ago, diaries are used in intensive care unit to limit these symptoms after a coma. In analogy, the diary for the patients with allogenic hematopoietic stem cell transplantation could be a mean to reduce the psychological adverse impact and long terms consequences. The investigators want to evaluate the psychological impact of a diary on the patients hospitalized for allogenic hematopoetic stem cell transplantation and on their relatives.

ELIGIBILITY:
Inclusion Criteria:

* patient age > 18 years
* patient hospitalized for an hematopoietic allogenic stem cell transplantation
* patient agreeing to participate

Exclusion Criteria:

* patient not hospitalized for an hematopoietic allogenic stem cell transplantation

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2019-11-01 (Actual); Primary Completion 2021-05-01 (Actual); Study Completion 2023-03-21 (Actual)

PRIMARY OUTCOMES:
Measure of diary impact on patient quality of life | at day 0
  the diary for patients with allogenic hematopoietic stem cell transplantation could be a mean to reduce the psychological adverse impact and long term consequences.
Measure of diary impact on patient quality of life | through the end of hospitalisation, an average of 3 weeks
  the diary for patients with allogenic hematopoietic stem cell transplantation could be a mean to reduce the psychological adverse impact and long term consequences.
Measure of diary impact on patient quality of life | at 30 days after transplantation
  the diary for patients with allogenic hematopoietic stem cell transplantation could be a mean to reduce the psychological adverse impact and long term consequences.
Measure of diary impact on patient quality of life | at day 100 after transplantation
  the diary for patients with allogenic hematopoietic stem cell transplantation could be a mean to reduce the psychological adverse impact and long term consequences.
Measure of diary impact on patient quality of life | 6 months after transplantation
  the diary for patients with allogenic hematopoietic stem cell transplantation could be a mean to reduce the psychological adverse impact and long term consequences.
Measure of diary impact on patient quality of life | a year after transplantation
  the diary for patients with allogenic hematopoietic stem cell transplantation could be a mean to reduce the psychological adverse impact and long term consequences.

SECONDARY OUTCOMES:
Measure of diary impact on health care team satisfaction | at day 0
  the diary for patients with allogenic hematopoietic stem cell transplantation could be a mean to reduce the psychological adverse impact and long term consequences.
Measure of diary impact on health care team satisfaction | through the end of hospitalisation, an average of 3 weeks
  the diary for patients with allogenic hematopoietic stem cell transplantation could be a mean to reduce the psychological adverse impact and long term consequences.
Measure of diary impact on health care team satisfaction | at 30 days after transplantation
  the diary for patients with allogenic hematopoietic stem cell transplantation could be a mean to reduce the psychological adverse impact and long term consequences.
Measure of diary impact on health care team satisfaction | at day 100 after transplantation
  the diary for patients with allogenic hematopoietic stem cell transplantation could be a mean to reduce the psychological adverse impact and long term consequences.
Measure of diary impact on health care team satisfaction | 6 months after transplantation
  the diary for patients with allogenic hematopoietic stem cell transplantation could be a mean to reduce the psychological adverse impact and long term consequences.
Measure of diary impact on health care team satisfaction | a year after transplantation
  the diary for patients with allogenic hematopoietic stem cell transplantation could be a mean to reduce the psychological adverse impact and long term consequences.
Measure of diary impact on patient relative quality of life | at day 0
  the diary for patients with allogenic hematopoietic stem cell transplantation could be a mean to reduce the psychological adverse impact and long term consequences.
Measure of diary impact on patient relative quality of life | through the end of hospitalisation, an average of 3 weeks
  the diary for patients with allogenic hematopoietic stem cell transplantation could be a mean to reduce the psychological adverse impact and long term consequences.
Measure of diary impact on patient relative quality of life | at 30 days after transplantation
  the diary for patients with allogenic hematopoietic stem cell transplantation could be a mean to reduce the psychological adverse impact and long term consequences.
Measure of diary impact on patient relative quality of life | at day 100 after transplantation
  the diary for patients with allogenic hematopoietic stem cell transplantation could be a mean to reduce the psychological adverse impact and long term consequences.
Measure of diary impact on patient relative quality of life | 6 months after transplantation
  the diary for patients with allogenic hematopoietic stem cell transplantation could be a mean to reduce the psychological adverse impact and long term consequences.
Measure of diary impact on patient relative quality of life | a year after transplantation
  the diary for patients with allogenic hematopoietic stem cell transplantation could be a mean to reduce the psychological adverse impact and long term consequences.

CONTACTS AND LOCATIONS:
Overall Officials: Delphine Lebon, MD, Principal Investigator — CHU Amiens; Marie Beaumont, MD, Principal Investigator — CHU Amiens
Locations (1):
- CHU Amiens, Amiens, France

IPD SHARING:
Plan to Share IPD: No